CLINICAL TRIAL: NCT02580461
Title: Renewing Caregiver Health and Well-being Through Exercise: A Randomized Controlled Trial
Brief Title: Renewing Caregiver Health and Well-being Through Exercise
Acronym: RECHARGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Nicole Culos-Reed, Professor, Faculty of Kinesiology,, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-2478
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Family Caregivers
Keywords: family caregivers; cancer; exercise intervention; center based
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Exercise Group (Experimental): One half of the participants enrolled in the 24 week center-based structured exercise and education program will be randomized to the immediate exercise group. The immediate exercise group will receive a 12 week center based structured exercise program followed by a 12 week maintenance of exercise program.
  Interventions: Behavioral: A 24 week center-based structured exercise and education program
- Delayed Exercise Group (No Intervention): One half of the participants enrolled in the 24 week center-based structured exercise and education program will be randomized to the delayed exercise group. This will be a wait list control group and the participants will receive no active intervention for 12 weeks. The wait list control group will then be enrolled in the 12 week structured exercise intervention.

INTERVENTIONS:
Behavioral: A 24 week center-based structured exercise and education program — The intervention will consist of a strength and aerobic exercise program. The exercise program will include twice weekly group resistance exercises classes, twice monthly group education classes, and individual activities to achieve 150 weekly minutes of aerobic activity. The resistance exercise and education classes will be run at a gym space at the University of Calgary. The wait-list control participants will be told not to change their activity levels throughout the 12 weeks of the trial. The wait list control participants will be enrolled into the exercise and education intervention once they have completed 12 weeks of wait-list control. A 12 week maintenance exercise program will be offered to all participants who finish the 12 week exercise and education program. The maintenance exercise program will consist of once weekly resistance group based exercise classes and individual activities to achieve 150 weekly minutes of aerobic physical activity.
  Arms: Immediate Exercise Group

SUMMARY:
The RECHARGE study is evaluating the effect of a 24 week structured exercise and education program on the physical and emotion health, quality of life, physical activity and fitness levels of family caregivers. Very little research has been done examining the impact of a structured exercise program designed for family caregivers of cancer patients. The purpose of this study is to determine if physical activity is effective in improving caregiver health and well-being.

DETAILED DESCRIPTION:
The REHCARGE study is a randomized control trial testing a structured exercise program for cancer family caregivers. One half of the participants enrolled will receive no exercise program until after twelve weeks have passed (the delayed start group) and the other half of the participants will start the exercise program right away. In addition to regular attendance at exercise classes, participants will also be asked to complete some measurements throughout the study including an initial assessment and one after 12 weeks and 24 weeks of the exercise programs. If participants are a part of the delayed start group, they will receive a fourth fitness assessment. Assessments include an evaluation of physical activity levels, quality of life, depression, sleep, and social support through survey type questionnaires as well as a fitness assessment to measure overall fitness and body composition. Participants will receive an individualized exercise program appropriate for their fitness level as well as 6 education sessions about healthy behaviors throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Currently providing physical care, instrumental or psychological support to an adult patient who has been diagnosed with any type of cancer.
* They must not have any physical health conditions that would restrict their participation in an aerobic and resistance exercise program.
* They must be willing to participate in two exercise classes per week at a gym space at the University of Calgary.
* They must not be planning on moving for the next 12 months
* Not currently meeting the Canadian Physical Activity Guidelines (150 minutes of aerobic activity per week and 2 sessions of resistance training per week) for the last three months.
* Be able to speak and read English

Exclusion Criteria:

* Providing care to a child with cancer Participants caring for a child with cancer will be excluded
* Participants with a health condition that limits their participation in a physical activity program will be excluded
* Participants who were previously caring for a cancer patient and that patient has now died (i.e. bereaved caregivers) will be excluded
* Participants meeting the Canadian Physical Activity guidelines for the past three months will be excluded
* Participants who cannot attend the group exercise classes will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 12 weeks
  The physical functioning score of the Medical Outcomes Short Form 36 will be the primary outcome

SECONDARY OUTCOMES:
Physical activity levels | 12 weeks
  Physical activity levels will be measured through standardized self-report questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary Health and Wellness Lab, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Cuthbert CA, King-Shier KM, Ruether JD, Tapp DM, Wytsma-Fisher K, Fung TS, Culos-Reed SN. The Effects of Exercise on Physical and Psychological Outcomes in Cancer Caregivers: Results From the RECHARGE Randomized Controlled Trial. Ann Behav Med. 2018 Jul 13;52(8):645-661. doi: 10.1093/abm/kax040. PMID 30010704
- [Derived] Cuthbert CA, King-Shier K, Tapp DM, Ruether D, Jackson C, Culos-Reed SN. Renewing caregiver health and wellbeing through exercise (RECHARGE): A randomized controlled trial. Contemp Clin Trials. 2016 Sep;50:273-83. doi: 10.1016/j.cct.2016.08.007. Epub 2016 Aug 13. PMID 27530087
- See also: Related Info — http://www.ucalgary.ca/healthandwellnesslab/